CLINICAL TRIAL: NCT06989489
Title: Design and Implementation of a Social Cognitive Theory-based Medication Adherence Intervention
Brief Title: Implementation of an Oral Chemotherapy Adherence Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LCCC2125-AIM3; K08CA279500 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-05-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Hematologic Malignancy
Keywords: oral anticancer agent; oral chemotherapy; adherence
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Surveys will be administered to two different groups, before implementation and after implementation of intervention.
Who Masked: Participant
Masking Description: Participants will not be aware that they are receiving a different follow up pattern from other patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care patients (No Intervention): Clinical pharmacists will follow their specific standards of procedure when educating patients on oral anticancer agents. No longitudinal following or tailored patient support will be provided. This group of participants will serve as the control group of the study.
- Intervention participants (Experimental): Participants enrolled in this adherence program will have individualized counseling sessions with their clinical pharmacists regarding their oral anticancer agent. Participants will be followed longitudinally and will receive tailored support.
  Interventions: Behavioral: Multilevel Adherence Intervention

INTERVENTIONS:
Behavioral: Multilevel Adherence Intervention — Participants enrolled in this adherence program will have individualized counseling sessions with their clinical pharmacists regarding their oral anticancer agent based on their risk-stratified monitoring category. Participants will be followed longitudinally and will receive tailored support.
  Other Names: Multicomponent Adherence Intervention
  Arms: Intervention participants

SUMMARY:
The goal of this study is to evaluate the effectiveness and usability of a newly developed oral anticancer agent adherence program implemented across 6 cancer clinics (two academic, two urban, and two rural). The study will include 160 adult participants with either solid tumors or hematologic malignancies who have been taking oral anticancer agents for at least six months.

This study will have two groups of participants, a pre- and post-implementation group. In the pre-implementation of the program group, investigators will administer a survey to the 80 participants and gather information about their medication prior to their enrollment of the program. Similarly, 80 participants who have been enrolled into this program for at least 6 months will serve as the post-implementation group. These patients will be administered the same survey. The results from both groups will be analyzed to see how effective the medication adherence program is.

DETAILED DESCRIPTION:
Participants enrolled in this adherence program will have individualized counseling sessions with their clinical pharmacists regarding their oral anticancer agent. The pharmacists will review with all their patients, information including proper administration, side effects, symptom management, and treatment plans. Participants will continue to have these counseling sessions with their pharmacists, until the patient becomes stable on the oral anticancer agent.

Once stable, the participant will be placed into one of three monitoring risk categories (low risk, medium risk, high risk), by the pharmacist, based on several factors. Each of the three monitor categories will have different monitoring intervals where patients will interact with the pharmacists differently. Additionally, each patient will have follow-up appointments and will have access to further education and will be reassessed each time. Furthermore, additional help will be provided to each patient based on their needs. Depending on the monitoring category, participants may meet with their pharmacist more and communicate either through electronic surveys or in-person visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥21 years-old) patients
* Diagnosed with a solid or hematologic malignancy
* Monotherapy on oral anticancer agent on treatment for at least 6 months

Exclusion criteria:

* Patients on time-limited or intermittent therapy (non-continuous)
* Patients on comfort (end-of-life) care
* Patients enrolled on hospice

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Oral Medication Adherence | Baseline and week 4
  Patient's medication adherence of their oral anticancer regiment will be quantified using the PROMIS- medication adherence Likert-type questionnaire, from strongly disagree to strongly agree. Score will change from 1 to 5, with a maximum of 50 and minimum of 10. A higher score reflects better adherence. These answers will help the investigators see if the program was effective in helping the patient's medication adherence.
Acceptability | After 6 months
  A study specific survey will be used to measure acceptability. Survey will have Likert-type questions, 1-5 strongly disagree to strongly agree, a higher score reflects better acceptance. Clinicians and administrators will answer the survey to capture their acceptability of the various aspects of the intervention.
Appropriateness | After 6 months
  A study specific survey will be used to measure appropriateness. Survey will have Likert-type questions, 1-5 strongly disagree to strongly agree, a higher score reflects better appropriateness. the survey will capture how well the clinicians and administrators graded the various aspects of the intervention.
Everyday use | After 6 months
  A study specific survey will be used to measure how applicable for everyday use. Survey will have Likert-type questions, 1-5 strongly disagree to strongly agree, a higher score reflects better everyday use. The survey will capture how easy the intervention is for clinicians and administrators.

SECONDARY OUTCOMES:
Medication knowledge | Baseline and 4 weeks
  A study specific survey that includes Likert-types and open-ended questions assessing the participant's knowledge on their medication and treatment will be used. Likert-style questions from strongly disagree to strongly agree with scores ranging from 1 to 5. Higher scores will reflect better knowledge of the participant's medication.
Patient perception | Baseline and 4 weeks
  A study specific survey that will include Likert-type questions assessing the participant's perceptions of their cancer care team will be used. Likert-style questions from strongly disagree to strongly agree with scores ranging from 1 to 5. Higher scores will reflect better perceptions of the participants cancer care provider, providers in general, and all people who work in healthcare.
Health literacy | Baseline and 4 weeks
  A study specific survey that will include Likert-type questions assessing the participant's health literacy of the instructions of their medication, treatment plan, healthcare professional explanations, and provider education will be used. Likert-style questions will range from not difficult to extremely difficult and scores ranging from 1 to 5. Higher scores will reflect stronger health literacy of the participants.
Self-efficacy | Baseline and 4 weeks
  A study specific survey will consist of multiple-choice questions regarding resources participants use to help them take their medications as well as a Likert-style question, from strongly disagree to strongly agree about how and when to call a pharmacist. Likert-style questions will have scores ranging from 1 to 5. Higher scores will reflect better self-efficacy of the participants.
Patient satisfaction | Baseline and 4 weeks
  A study specific survey will consist of Likert-style questions, ranging from strongly disagree to strongly agree, regarding the participant's satisfaction of their healthcare team, pharmacy team, care coordination, treatment plan, and education received since starting treatment will be used. Likert-style questions will have scores ranging from 1 to 5. Higher scores will reflect stronger satisfaction of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Benyam Muluneh, PharmD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials